CLINICAL TRIAL: NCT01126346
Title: HOPE Program: Quality of Life Enhancement and Survivorship Care
Brief Title: Quality of Life and Survivorship Care in Patients Undergoing Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00013172; NCI-2010-00980; CCCWFU 97110 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-05-13; First posted 2010-05-19 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Advanced Malignant Mesothelioma; Carcinoma of the Appendix; Ovarian Sarcoma; Ovarian Stromal Cancer; Pseudomyxoma Peritonei; Recurrent Colon Cancer; Recurrent Malignant Mesothelioma; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Stage III Colon Cancer; Stage III Ovarian Epithelial Cancer; Stage III Ovarian Germ Cell Tumor; Stage IV Colon Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Appendiceal Neoplasms; Pseudomyxoma Peritonei; Colonic Neoplasms; Mesothelioma, Malignant; Carcinoma, Ovarian Epithelial | interventions — Referral and Consultation; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm I (Experimental): Patients and their caregiver(s) receive a hyperthermic intraperitoneal chemotherapy (HIPEC) orientation with a Survivorship Navigator (SN) over 90 minutes following their initial surgical consult. Patients then receive telephone calls over 20-30 minutes from the SN once weekly for 3 weeks prior to HIPEC. After HIPEC, patients meet with the SN for 20-30 minutes to discuss adjustments and adaptation to the surgery and hospitalization 3-4 days post-HIPEC, biweekly for two weeks and weekly thereafter until hospital discharge. After hospital discharge, patients receive telephone calls from the SN twice monthly for 1 month.
  Interventions: Behavioral: HIPEC Orientation; Behavioral: Consultation with Survivorship Navigator; Other: Questionnaires

INTERVENTIONS:
Behavioral: HIPEC Orientation — Introduction to SRB (survivorship resource book); Clinic Tour; Lunch with Question and Answer Session
  Other Names: orientation
Behavioral: Consultation with Survivorship Navigator — Weekly psychosocial support via phone from Survivorship Navigator for 3 weeks prior to HIPEC; Inpatient consults occurring 3 to 4 days post-HIPEC and biweekly for 2 weeks and weekly until hospital discharge; Post-Hospital Discharge consults via phone twice per month for one month
  Other Names: Consultation
Other: Questionnaires — Questionnaires Completed at 4 time points: T1 pre-HIPEC orientation, T2 with in 1 week of orientation, T3 1 month post HIPEC and T4 3 months post HIPEC. Questionnaires include Utility of SRB, Medical Outcomes Study Health Survey, Short Form (SF-12), Center for Epidemiologic Studies-Depression Scale (CES-D), The Brief Illness Perception Questionnaire, The Distress Thermometer, The State-Trait Anxiety Inventory (STAI)

SUMMARY:
RATIONALE: An orientation and patient education program and telephone counseling may help improve the quality of life in patients with peritoneal surface malignancies.

PURPOSE: This clinical trial studies quality of life and survivorship care in patients undergoing surgery and chemotherapy for peritoneal surface malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess feasibility of instituting an orientation program, brief follow up care and phone calls in this patient population.

SECONDARY OBJECTIVES:

I. Reduce pre-treatment distress and anxiety. II. Improve pre-treatment self-efficacy. III. Provide educational material delivered by the SRB. IV. Improve overall post-operative QOL ratings at 3 months, relative to discharge.

OUTLINE:

Patients and their caregiver(s) receive a hyperthermic intraperitoneal chemotherapy (HIPEC) orientation with a Survivorship Navigator (SN) over 90 minutes following their initial surgical consult. Patients then receive telephone calls over 20-30 minutes from the SN once weekly for 3 weeks prior to HIPEC. . After HIPEC, patients meet with the SN for 20-30 minutes to discuss adjustments and adaptation to the surgery and hospitalization 3-4 days post-HIPEC, biweekly for two weeks, and weekly thereafter until hospital discharge. After hospital discharge, patients receive telephone calls from the SN twice monthly for 1 month.

ELIGIBILITY:
Inclusion

* Patients who undergo CS and HIPEC for peritoneal surface malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Assess feasibility of instituting an orientation program, brief follow up care and phone calls in this patient population | Baseline to 3 months post discharge
  Utility of SRB, Medical Outcomes Study Health Survey, Short Form (SF-12), Center for Epidemiologic Studies-Depression Scale (CES-D), The Brief Illness Perception Questionnaire, The Distress Thermometer, The State-Trait Anxiety Inventory (STAI)

SECONDARY OUTCOMES:
Reduce pre-treatment distress and anxiety | Pre-HIPEC to Day 0
  Compared t-tests will be conducted for the CESD and STAI (state anxiety subscale).
Improve pre-treatment self-efficacy | Pre-HIPEC to Day 0
  Mean scores on the distress thermometer will be compared as well as individual patient changes.
Provide educational material delivered by the SRB | Pre-HIPEC to Day 0
  Form to assess utility of the Survivorship Resource Book
Improve overall post-operative QOL ratings at 3 months, relative to discharge | 3 months post discharge
  Improve post-operative QOL ratings at 3 months, relative to discharge. Repeated measures analysis of covariance (ANCOVA) will be utilized with the FACT scales.

CONTACTS AND LOCATIONS:
Overall Officials: Richard McQuellon, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States